CLINICAL TRIAL: NCT06330441
Title: Pancreatic Cancer Screening in a Population at High Risk
Acronym: ScrePan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk Memorial Cancer Institute (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MOU-2021-01
Record Dates: First submitted 2023-12-31; First posted 2024-03-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Hereditary Diseases; Pancreatitis, Chronic
Keywords: pancreatic ductal adenocarcinoma; screening programme; high-risk population
MeSH Terms: conditions — Genetic Diseases, Inborn; Pancreatitis, Chronic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A - chronic pancreatitis (Experimental): Chronic pancreatitis, due to cystic fibrosis
  Interventions: Procedure: endoscopic ultrasonography; Procedure: magnetic resonance; Diagnostic Test: laboratory examination
- B1 - genetic predisposition (STK11, CDKN2A, PRSS1) (Experimental): Persons with a confirmed diagnosis of Peutz-Jeghers syndrome (STK11 mutation) or familial melanoma syndrome (CDKN2A mutation), hereditary pancreatitis (PRSS1 mutation)
  Interventions: Procedure: endoscopic ultrasonography; Procedure: magnetic resonance; Diagnostic Test: laboratory examination
- B2 - genetic predisposition of hereditary syndromes (Experimental): Persons with a confirmed diagnosis of hereditary syndromes and at the same time with the condition of at least one relative of the first or second degree with a diagnosis of pancreatic ductal adenocarcinoma in family anamnesis; i.e. Lynch syndrome (mut: MLH1, MSH2, MSH6 a PMS2, EPCAM), HBOC (mut: BRCA1, BRCA2, PALB2, ATM), familial adenomatous polyposis (mut: APC), Li-Fraumeni syndrome (mut: TP53)
  Interventions: Procedure: endoscopic ultrasonography; Procedure: magnetic resonance; Diagnostic Test: laboratory examination
- C - positive family anamnesis (Experimental): Persons with positive family anamnesis of pancreatic ductal adenocarcinoma without proven hereditary syndrome
  Interventions: Procedure: endoscopic ultrasonography; Procedure: magnetic resonance; Diagnostic Test: laboratory examination

INTERVENTIONS:
Procedure: endoscopic ultrasonography — endoscopic ultrasonography - frequency defined by arm
  Other Names: EUS
Procedure: magnetic resonance — magnetic resonance - frequency defined by arm
  Other Names: MR
Diagnostic Test: laboratory examination — hematology, biochemistry, Na+, K+, Cl-, Ca2+, bilirubin, ALT, AST, GGT, ALP, lactate dehydrogenase, creatinine, urea, fasting glycemia, HbA1c, alpha-amylase, LPS, albumin, total protein, CA19-9, CEA
  Other Names: LAB

SUMMARY:
Pancreatic cancer is one of the diseases with the worst prognosis, which is mainly due to the initial asymptomatic prognosis. Unfortunately, the incidence of this disease in the Czech Republic is still increasing. In a certain proportion of patients, it is possible to predict the disease, e.g. due to family burdens. Regular follow-up of such individuals is the subject of the SCREPAN study: "Pancreatic Cancer Screening in High-Risk Persons".

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the cancers with the worst prognosis. Mortality in this disease is almost equal to the incidence. In the Czech Republic, the incidence of this cancer has an upward trend, in 2017, 21.2 new cases per 100,000 people were reported, which represents a more than double increase compared to the data from the 1970s.

Pancreatic cancer is associated with an extremely poor prognosis for several reasons. It is usually diagnosed at an advanced stage, which is often due to the asymptomatic course of the disease or non-specific symptoms, the lack of sensitive and specific tumor markers, and difficult diagnosis by imaging methods in the early stages. Five-year survival, regardless of clinical stage, is between 7-9%.

Resectable disease is diagnosed in only 10% of patients, in which the 5-year survival rate is 37 %, locally advanced unresectable disease is detected in about 30 % of patients with a 5-year survival of 12 %, and metastatic disease is found in about 60 % of patients, with a 5-year survival rate of only around 3 %.

The poor prognosis of this disease is also due to the limited possibilities of screening and curative intervention for a short "lead time" in rapidly metastatic disease.

Pancreatic cancer screening is not suitable for the non-selected population. On the contrary, it is important for individuals with a high risk of developing this disease. In these subjects, early diagnosis during screening demonstrated a higher number of curative resections and longer survival.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study
* age 18+
* arms specific criteria:

A:

* chronic pancreatic disease in the context of cystic fibrosis or chronic pancreatitis
* age 50+

B1:

* confirmed Peutz-Jegherson syndrome (mutSTK11) + age over 35 years or 10 years earlier than pancreatic ductal adenocarcinoma was diagnosed in the youngest family member
* familial melanoma syndrome (mutCDKN2A) + age over 40 years or 10 years before pancreatic ductal adenocarcinoma was diagnosed in the youngest family member
* confirmed hereditary pancreatitis (mutPRSS1) + age over 40 years or 20 years after the first attack

B2:

* confirmed diagnosis of hereditary syndrome (Lynch syndrome /mutMLH1, mutMSH2, mutMSH6, mutPMS2, mutEPCAM/, HBOC /mutBRCA1, mutBRCA2, mutPALB2, mutATM/, familial adenomatous polyposis /mutAPC/, Li-Fraumeni syndrome /mutTP53/)
* at least one relative with a diagnosis of pancreatic ductal adenocarcinoma in family anamnesis at the same time (Grade I or II relative)
* age over 50 years, or 10 years before the pancreatic ductal adenocarcinoma was diagnosed in the youngest relative - which comes first

C:

* positive family anamnesis of pancreatic ductal adenocarcinoma without hereditary syndrome context
* age 50+ or 10 years earlier than the youngest relative with pancreatic ductal adenocarcinoma - screening is recommended for all first-degree relatives of affected family members

Exclusion Criteria:

* Inability to undergo radical curative surgery for a pancreatic tumor.
* Inability to undergo scheduled imaging examinations.
* Incurable malignant cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-01-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with newly diagnosed pancreatic ductal adenocarcinoma | From date of subject enrollment annualy in determined examinations according to the protocol schedule until the date of PDAC diagnosis or up to 60 months of subject participation in the study
  Number of participants (in risk population) with newly diagnosed pancreatic cancer

SECONDARY OUTCOMES:
Methods yield comparison | through study completion, an average of 1 year
  Comparison of magnetic resonance versus endoscopic ultrasonography yield
Screening methods cost-effectiveness | through study completion, an average of 1 year
  Comparison of magnetic resonance versus endoscopic ultrasonography cost effectiveness
KRAS mutation status evaluation | From the date of subject enrollment annualy in determined examinations according to the protocol schedule until the date of PDAC diagnosis or up to 60 months of subject participation in the study
  KRAS mutation status defined by number of positive droplets on drop digital PCR using material from liquid biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Canto MI, Harinck F, Hruban RH, Offerhaus GJ, Poley JW, Kamel I, Nio Y, Schulick RS, Bassi C, Kluijt I, Levy MJ, Chak A, Fockens P, Goggins M, Bruno M; International Cancer of Pancreas Screening (CAPS) Consortium. International Cancer of the Pancreas Screening (CAPS) Consortium summit on the management of patients with increased risk for familial pancreatic cancer. Gut. 2013 Mar;62(3):339-47. doi: 10.1136/gutjnl-2012-303108. Epub 2012 Nov 7. PMID 23135763
- [Background] Syngal S, Brand RE, Church JM, Giardiello FM, Hampel HL, Burt RW; American College of Gastroenterology. ACG clinical guideline: Genetic testing and management of hereditary gastrointestinal cancer syndromes. Am J Gastroenterol. 2015 Feb;110(2):223-62; quiz 263. doi: 10.1038/ajg.2014.435. Epub 2015 Feb 3. PMID 25645574
- [Background] Stoffel EM, McKernin SE, Brand R, Canto M, Goggins M, Moravek C, Nagarajan A, Petersen GM, Simeone DM, Yurgelun M, Khorana AA. Evaluating Susceptibility to Pancreatic Cancer: ASCO Provisional Clinical Opinion. J Clin Oncol. 2019 Jan 10;37(2):153-164. doi: 10.1200/JCO.18.01489. Epub 2018 Nov 20. PMID 30457921
- [Background] Abe T, Blackford AL, Tamura K, Ford M, McCormick P, Chuidian M, Almario JA, Borges M, Lennon AM, Shin EJ, Klein AP, Hruban RH, Canto MI, Goggins M. Deleterious Germline Mutations Are a Risk Factor for Neoplastic Progression Among High-Risk Individuals Undergoing Pancreatic Surveillance. J Clin Oncol. 2019 May 1;37(13):1070-1080. doi: 10.1200/JCO.18.01512. Epub 2019 Mar 18. PMID 30883245
- [Background] Bartsch DK, Slater EP, Carrato A, Ibrahim IS, Guillen-Ponce C, Vasen HF, Matthai E, Earl J, Jendryschek FS, Figiel J, Steinkamp M, Ramaswamy A, Vazquez-Sequeiros E, Munoz-Beltran M, Montans J, Mocci E, Bonsing BA, Wasser M, Kloppel G, Langer P, Fendrich V, Gress TM. Refinement of screening for familial pancreatic cancer. Gut. 2016 Aug;65(8):1314-21. doi: 10.1136/gutjnl-2015-311098. Epub 2016 May 24. PMID 27222532
- [Background] Harinck F, Konings IC, Kluijt I, Poley JW, van Hooft JE, van Dullemen HM, Nio CY, Krak NC, Hermans JJ, Aalfs CM, Wagner A, Sijmons RH, Biermann K, van Eijck CH, Gouma DJ, Dijkgraaf MG, Fockens P, Bruno MJ; Dutch research group on pancreatic cancer surveillance in high-risk individuals. A multicentre comparative prospective blinded analysis of EUS and MRI for screening of pancreatic cancer in high-risk individuals. Gut. 2016 Sep;65(9):1505-13. doi: 10.1136/gutjnl-2014-308008. Epub 2015 May 18. PMID 25986944
- [Background] Corral JE, Das A, Bruno MJ, Wallace MB. Cost-effectiveness of Pancreatic Cancer Surveillance in High-Risk Individuals: An Economic Analysis. Pancreas. 2019 Apr;48(4):526-536. doi: 10.1097/MPA.0000000000001268. PMID 30946242
- [Background] Vasen H, Ibrahim I, Ponce CG, Slater EP, Matthai E, Carrato A, Earl J, Robbers K, van Mil AM, Potjer T, Bonsing BA, de Vos Tot Nederveen Cappel WH, Bergman W, Wasser M, Morreau H, Kloppel G, Schicker C, Steinkamp M, Figiel J, Esposito I, Mocci E, Vazquez-Sequeiros E, Sanjuanbenito A, Munoz-Beltran M, Montans J, Langer P, Fendrich V, Bartsch DK. Benefit of Surveillance for Pancreatic Cancer in High-Risk Individuals: Outcome of Long-Term Prospective Follow-Up Studies From Three European Expert Centers. J Clin Oncol. 2016 Jun 10;34(17):2010-9. doi: 10.1200/JCO.2015.64.0730. Epub 2016 Apr 25. PMID 27114589
- [Background] Canto MI, Almario JA, Schulick RD, Yeo CJ, Klein A, Blackford A, Shin EJ, Sanyal A, Yenokyan G, Lennon AM, Kamel IR, Fishman EK, Wolfgang C, Weiss M, Hruban RH, Goggins M. Risk of Neoplastic Progression in Individuals at High Risk for Pancreatic Cancer Undergoing Long-term Surveillance. Gastroenterology. 2018 Sep;155(3):740-751.e2. doi: 10.1053/j.gastro.2018.05.035. Epub 2018 May 24. PMID 29803839
- [Background] Dbouk M, Katona BW, Brand RE, Chak A, Syngal S, Farrell JJ, Kastrinos F, Stoffel EM, Blackford AL, Rustgi AK, Dudley B, Lee LS, Chhoda A, Kwon R, Ginsberg GG, Klein AP, Kamel I, Hruban RH, He J, Shin EJ, Lennon AM, Canto MI, Goggins M. The Multicenter Cancer of Pancreas Screening Study: Impact on Stage and Survival. J Clin Oncol. 2022 Oct 1;40(28):3257-3266. doi: 10.1200/JCO.22.00298. Epub 2022 Jun 15. PMID 35704792
- [Background] Sawhney MS, Calderwood AH, Thosani NC, Rebbeck TR, Wani S, Canto MI, Fishman DS, Golan T, Hidalgo M, Kwon RS, Riegert-Johnson DL, Sahani DV, Stoffel EM, Vollmer CM Jr, Qumseya BJ; Prepared by: ASGE STANDARDS OF PRACTICE COMMITTEE. ASGE guideline on screening for pancreatic cancer in individuals with genetic susceptibility: summary and recommendations. Gastrointest Endosc. 2022 May;95(5):817-826. doi: 10.1016/j.gie.2021.12.001. Epub 2022 Feb 16. No abstract available. PMID 35183358